CLINICAL TRIAL: NCT07388459
Title: Natural History, Evolution, and Clinical Features of Autoimmune Atrophic Gastritis
Acronym: NH-GAA
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Emanuela Miceli, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: NH-GAA
Record Dates: First submitted 2025-03-19; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-02

CONDITIONS: Atrophic Gastritis
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Complete cell blood count, serum gastrin and chromogranin A levels, vitamin B12, folate, homocysteine iron balance, PCA, serum levels of calcium, 1,25(OH)2-vitamin D, 25(OH)-vitamin D, parathyroid hormone (PTH), TSH reflex, phosphate and auto-antibodies (TPO, TG, TSH receptor, transglutaminase) will be evaluated once a year. In a subset of 80 randomly selected AAG patients (only patient enrolled at Fondazione IRCCS Policlinico San Matteo, S. C. General Medicina I), with an age range of 30-65, with a M:F ratio of 1:1 serum markers of bone turnover as, osteoprotegerin (OPG), Receptor Antagonist of NF-kB Ligand (RANKL), COOH-terminal propeptide of type I procollagen (propeptide), IL-17, IL-15, IL-21 will be evaluated only once. Stool samples for microbiome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- We enroll all atrophic gastritis diagnosis is made according to the updated Sydney System criteria

SUMMARY:
Autoimmune atrophic gastritis (AAG) is an immune-mediated disorder characterized by the loss of oxyntic glands and mucosal atrophy1.Specific autoantibodies directed to gastric parietal cells (PCA) and/or to intrinsic factors are inconstantly present1.Despite its morbidity, data on the epidemiology are scant. Its global prevalence has been estimated to be 0.5-4.5%.Hypo-achlorhydria and lack of intrinsic factor lead to malabsorption of many nutrients, as vit. B12, iron and calcium.A damage on elevated turnover cells may develop, affecting hemopoiesis, nervous system, gut, and myocardium, depicting a systemic disease.Moreover, one of the primary function of gastric acidity as a bactericidal defensive barrier is impaired resulting in both gastric and intestinal microbiota modification. It was recently shown that conditions causing hypo-achlorhydria modify the composition of microbiota from stomach to colon. In particular, at colonic level a decrease in the abundance of commensal bacteria associated to a reduction in microbial diversity and an increase of oral bacteria in the stool were shown.The clinical spectrum is unspecific, especially in early stages, leading to substantial diagnostic delay.Patients may be asymptomatic or complain of gastrointestinal manifestations such as atrophic glossitis, malabsorption, diarrhea, and dyspepsia.These symptoms are insufficient for the diagnosis.Neurological and psychiatric symptoms are often overlooked; myocardial infarction due to demand imbalance may occur.Most of AAG manifestations and complications are due to cyanocobalamin deficiency that may be clinically silent for years.Vit. B12 deficiency has also been associated with infertility, very early recurrent miscarriage, failure of assisted reproductive technologies, and neural tube defects.Furthermore, AAG is a preneoplastic condition as may predispose to the development of type I carcinoids and gastric adenocarcinoma.A previous publication of our group on the NH of AAG,showed that all patients evolved into a higher degree of gastric atrophy and/or metaplasia; additionally,6.3%of these patients developed a neoplastic complication (median time of 3 yo).These data underlined the need to feel the gap of knowledge in the identification and characterization of the factors promoting neoplastic development or associated with carcinogenesis.Moreover, strategies for prevention and management of non-neoplastic complications and extra-gastrointestinal manifestation have to be better determined Hence, a larger, prospective study looking at this issue is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥18 years;
* AAG diagnosis is made according to the updated Sydney System criteria referring to a tertiary outpatient clinic dedicated;
* Signed written informed consent.

Exclusion Criteria:

* Patients with uncertain histopathological findings;
* Patients with persistent or active Helicobacter pylori infection;
* Patients with long-term proton pump inhibitor users and atrophic pangastritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both genders aged ≥ 18 years with atrophic gastritis being treated at Fondazione IRCCS Policlinico San Matteo
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clarify the natural history and the epidemiology of AAG in order to early diagnose patients, and to prevent irreversible complications | Baseline visit: all patients will be evaluated and all laboratory test required for protocol will be performed. 6 months, patients will be evaluated, for symptoms associated to AAG with VAS scale. 12 months a last evaluation will be performed.
  * The incidence of oncological gastric complications occurring in all autoimmune gastritis patients (potential, mild, moderate, severe)
  * The correlates of oncological complications, including laboratory markers, family history, autoimmune comorbidities, clinical features, so to identify clinical clusters and cluster-specific correlate.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Medicina Generale 1, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No